CLINICAL TRIAL: NCT04118010
Title: Vitamin D and Prebiotics for Intestinal Health in Cystic Fibrosis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Vin Tangpricha, Principal Investigator, Emory University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB00114230
Record Dates: First submitted 2019-10-04; First posted 2019-10-07 (Actual); Results first posted 2024-02-07 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-01

CONDITIONS: Cystic Fibrosis; Dysbiosis
Keywords: Cystic Fibrosis; Gastrointestinal Dysbiosis; Vitamin D; Prebiotic; Inulin; Gut microbiome; Intestinal inflammation; Intestinal absorption
MeSH Terms: conditions — Cystic Fibrosis; Dysbiosis | interventions — Cholecalciferol; Inulin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Vitamin D3 and Inulin (Active Comparator): Vitamin D3 50,000 IU/week and 12 g/day chicory-derived prebiotic inulin for 12 weeks
  Interventions: Drug: Vitamin D3; Drug: Inulin
- Vitamin D3 and placebo Inulin (Active Comparator): Vitamin D3 50,000 IU/week and 12 g/day corn-derived maltodextrin/day as the prebiotic placebo for 12 weeks
  Interventions: Drug: Vitamin D3; Drug: Placebo Inulin
- Placebo vitamin D3 and Inulin (Active Comparator): Matching to Vitamin D3 placebo capsules, and 12 g/day chicory-derived prebiotic inulin for 12 weeks
  Interventions: Drug: Placebo vitamin D3; Drug: Inulin
- Placebo vitamin D3 and placebo Inulin (Placebo Comparator): Matching to Vitamin D3 placebo capsules, and 12 g/day corn-derived maltodextrin/day as the prebiotic placebo for 12 weeks
  Interventions: Drug: Placebo vitamin D3; Drug: Placebo Inulin

INTERVENTIONS:
Drug: Vitamin D3 — High-dose vitamin D3 50,000 IU /week for 12 weeks
  Arms: Vitamin D3 and Inulin; Vitamin D3 and placebo Inulin
Drug: Placebo vitamin D3 — Matching to Vitamin D3 placebo capsules for 12 weeks
  Arms: Placebo vitamin D3 and Inulin; Placebo vitamin D3 and placebo Inulin
Drug: Inulin — Chicory-derived prebiotic inulin 12 g/day for 12 weeks
  Arms: Placebo vitamin D3 and Inulin; Vitamin D3 and Inulin
Drug: Placebo Inulin — Corn-derived maltodextrin 12g/day as the prebiotic placebo for 12 weeks
  Arms: Placebo vitamin D3 and placebo Inulin; Vitamin D3 and placebo Inulin

SUMMARY:
The study will assess if administration of high-dose vitamin D and a commonly used prebiotic (inulin) is effective to reduce gastrointestinal dysbiosis and to improve critical intestinal functions in Cystic Fibrosis with the additive or synergistic effects of the combination of vitamin D + inulin.

DETAILED DESCRIPTION:
Cystic fibrosis (CF) is the most common life-shortening genetic condition among Caucasians in the United States. Individuals with CF have an altered gastrointestinal (GI) microbiota, which may be a result of chronic systemic inflammation and infection, frequent use of antibiotics, and/or medically prescribed and habitual high-fat/high-calorie diets.

The study will assess if administration of high-dose vitamin D and a commonly used prebiotic (inulin) is effective to reduce gastrointestinal dysbiosis and to improve critical intestinal functions in Cystic Fibrosis.

ELIGIBILITY:
Inclusion Criteria:

1. male and female patients (age > 18 years) with confirmed CF by genetic mutation and/or sweat chloride testing,
2. not currently on oral or systemic antibiotics for pulmonary exacerbation,
3. vitamin D deficient/insufficient (25(OH)D, 6 - 30 ng/mL) with most recent 25(OH)D in the past 12 months,
4. use of CFTR modulator therapy is allowed

Exclusion Criteria:

1. severe vitamin D deficiency 25(OH)D ≤ 5 ng/mL or hypocalcemia or hypercalcemia,
2. active GI disease, abdominal pain and/or diarrhea,
3. chronic kidney disease worse than stage 3 (eGFR < ml/min per 1.73 m2),
4. any vitamin D supplement use >2,000 IU or vitamin D analogue (patients who are taking more than 2,000 IU of vitamin D must agree to stop the vitamin D for 6 weeks and take less than 2,000 IU of vitamin D during the study),
5. use of immunosuppressants or history of organ transplantation,
6. current use of probiotics or prebiotics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-03-13 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vin Tangpricha, MD, Principal Investigator — Emory University
Locations (1):
- Emory Clinic, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual de-identified participant data (including data dictionaries) be shared with listed investigators
Supporting Information: Study Protocol, SAP
Time Frame: Projected December 2023
Access Criteria: Protocol and reported primary and secondary outcomes will be be shared on request for statistical analyses with listed investigators

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Vitamin D3 and Inulin | Vitamin D3 and Placebo Inulin | Placebo Vitamin D3 and Inulin | Placebo Vitamin D3 and Placebo Inulin
Started | 10 | 10 | 10 | 10
Completed | 7 | 8 | 7 | 9
Not Completed | 3 | 2 | 3 | 1

BASELINE CHARACTERISTICS:
Population: Patients analyzed include participants that completed the trial.
Groups:
- Total: Total of all reporting groups
Arm/Group | Vitamin D3 and Inulin | Vitamin D3 and Placebo Inulin | Placebo Vitamin D3 and Inulin | Placebo Vitamin D3 and Placebo Inulin | Total
Number analyzed (Participants) | 7 | 8 | 7 | 9 | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.3 (5.4) | 29.3 (7.9) | 39.6 (15.6) | 34.4 (14.2) | 33.1 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 5 | 4 | 13
  Male | 6 | 5 | 2 | 5 | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 7 | 8 | 7 | 7 | 29
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 2 | 2
Region of Enrollment [Number; unit: participants]
  United States | 7 | 8 | 7 | 9 | 31

OUTCOME MEASURES:

1. Primary Outcome: Shannon Index
Description: The Shannon Index is a measure of diversity of microbial species that takes into account both abundance (the number of species present) and evenness (how close the numbers for each species are). The Shannon index can be calculated using the following equation: H= -∑(i=1)^s pi ln(pi). A value of zero for H indicates that a community has only one species. The higher the value of H, the higher the diversity of species in a particular community.
  Sputum microbiota analysis was measured using this ecological diversity measure. Sputum samples were collected via a sputum kit.
Time Frame: Baseline, 12 weeks post-intervention
Measure: Mean (Standard Deviation); unit: Shannon index
Arm/Group | Vitamin D3 and Inulin | Vitamin D3 and Placebo Inulin | Placebo Vitamin D3 and Inulin | Placebo Vitamin D3 and Placebo Inulin
Number analyzed (Participants) | 7 | 8 | 7 | 9
Shannon index
  Baseline | 5.02 (0.392) | 4.96 (0.165) | 5.28 (0.196) | 5.73 (0.081)
  12 weeks post-intervention | 5.02 (0.392) | 5.05 (0.169) | 5.24 (0.229) | 5.41 (0.097)

2. Primary Outcome: Change in Species Richness Index From Baseline
Description: Stool microbiota analysis will be measured using this ecological diversity measure. Stool samples will be collected using a stool kit provided to the participant.
Time Frame: Baseline, 12 weeks post-intervention
Population: Stool and serum samples were not collected due to Emory operations being disrupted due to COVID pandemic.
Arm/Group | Vitamin D3 and Inulin | Vitamin D3 and Placebo Inulin | Placebo Vitamin D3 and Inulin | Placebo Vitamin D3 and Placebo Inulin
Number analyzed (Participants) | 0 | 0 | 0 | 0

3. Secondary Outcome: Change in GI Microbiota Diversity
Description: Changes in GI microbiota diversity will be determined using 16S rRNA gene sequencing and microbiome-dependent metabolites pathways in stool and plasma using high-resolution metabolomics analysis.Changes in GI microbiota diversity will be reported as the Shannon Index.
Time Frame: Baseline, 12 weeks post-intervention
Population: Stool and serum samples were not collected due to Emory operations being disrupted due to COVID pandemic.
Arm/Group | Vitamin D3 and Inulin | Vitamin D3 and Placebo Inulin | Placebo Vitamin D3 and Inulin | Placebo Vitamin D3 and Placebo Inulin
Number analyzed (Participants) | 0 | 0 | 0 | 0

4. Secondary Outcome: Change in GI Microbiota Richness
Description: Changes in GI microbiota richness will be determined using 16S rRNA gene sequencing and microbiome-dependent metabolites pathways in stool and plasma using high-resolution metabolomics analysis.Changes in GI microbiota richness will be reported as a number of populations of microorganisms.
Time Frame: Baseline, 12 weeks post-intervention
Population: Stool and serum samples were not collected due to Emory operations being disrupted due to COVID pandemic.
Arm/Group | Vitamin D3 and Inulin | Vitamin D3 and Placebo Inulin | Placebo Vitamin D3 and Inulin | Placebo Vitamin D3 and Placebo Inulin
Number analyzed (Participants) | 0 | 0 | 0 | 0

5. Secondary Outcome: Change in GI Microbiota Composition
Description: Changes in GI microbiota composition will be determined using 16S rRNA gene sequencing and microbiome-dependent metabolites pathways in stool and plasma using high-resolution metabolomics analysis.Changes in GI microbiota composition will be reported as a percentage of bacteria.
Time Frame: Baseline, 12 weeks post-intervention
Population: Stool and serum samples were not collected due to Emory operations being disrupted due to COVID pandemic.
Arm/Group | Vitamin D3 and Inulin | Vitamin D3 and Placebo Inulin | Placebo Vitamin D3 and Inulin | Placebo Vitamin D3 and Placebo Inulin
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Information on adverse events was collected beginning at the baseline assessment and continued through the final assessment at Week 12.
Arm/Group | Vitamin D3 and Inulin | Vitamin D3 and Placebo Inulin | Placebo Vitamin D3 and Inulin | Placebo Vitamin D3 and Placebo Inulin
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/8 | 0/7 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/8 | 0/7 | 0/9
Other Adverse Events (participants affected / at risk) | 0/7 | 0/8 | 0/7 | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-10-31): https://cdn.clinicaltrials.gov/large-docs/10/NCT04118010/Prot_SAP_000.pdf